CLINICAL TRIAL: NCT01355159
Title: Effect of Folic Acid Supplementation in Pregnancy on Preeclampsia-Folic Acid Clinical Trial (FACT)
Brief Title: High Dose Folic Acid Supplementation Throughout Pregnancy for Preeclampsia Prevention
Acronym: FACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2009-107; ISRCTN23781770 (Other: controlled-trials.com)
Record Dates: First submitted 2011-05-11; First posted 2011-05-17 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Pregnancy Complications; Preeclampsia
Keywords: Pregnancy; Folic Acid supplementation; Preeclampsia
MeSH Terms: conditions — Pregnancy Complications; Pre-Eclampsia | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Folic Acid 4 mg (Experimental): Folic Acid 1.0 mg x 4 tablets will be taken daily by oral administration. The majority of women in the study will routinely take 1.0 mg folic acid in a prenatal vitamin supplement, as recommended by their primary obstetrical provider; the study requirements do not require that participants change their practice. Therefore the actual total daily dose may be up to 5.1 mg of folic acid
  Interventions: Drug: Folic Acid 4 mg
- Placebo (Placebo Comparator): Women will be randomised in a 1:1 ratio to folic acid 4.0 mg or placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Folic Acid 4 mg — Folic Acid 1.0 mg or placebo x 4 tablets will be taken daily by oral administration. The majority of women in the study will routinely take 1.0 mg folic acid in a prenatal vitamin supplement, as recommended by their primary obstetrical provider; the study requirements do not require that participants change their practice. Therefore the actual total daily dose may be up to 5.1 mg of folic acid
  Other Names: Folate
  Arms: Folic Acid 4 mg
Drug: Placebo — Placebo x 4 tablets will be taken daily by oral administration.
  Arms: Placebo

SUMMARY:
To determine the efficacy of high dose folic acid supplementation for prevention of preeclampsia in women with at least one risk factor: pre-existing hypertension, pre-pregnancy diabetes (type 1 or 2), twin pregnancy, preeclampsia in a previous pregnancy, or body mass index ≥35. It was hypothesized that high dose (4.0 mg per day) supplementation starting in early pregnancy and continued throughout the entire pregnancy will lower the incidence of preeclampsia in pregnant women at high risk of developing preeclampsia.

DETAILED DESCRIPTION:
Preeclampsia is a complication of pregnancy which affects at least 5% of all pregnancies worldwide and has serious health consequences to these women and their babies. Preeclampsia is hypertension (high blood pressure) in pregnancy with proteinuria. Proteinuria is when protein is found in the urine, and it is a sign that the kidneys are not functioning properly. The only effective treatment for preeclampsia is delivery of the baby. Because delivery may be required before the anticipated date of delivery; preeclampsia is also one of the leading causes of preterm delivery and accounts for 25% of very low birth weight infants. Recent research has also shown that women who have had preeclampsia during pregnancy are more likely to be at risk for future cardiovascular events later in life.

Recently some studies have shown that supplementation with multivitamins containing folic acid is associated with a reduced risk of developing preeclampsia. These findings also suggested that for the prevention of preeclampsia, a high dose of folic acid (much higher than the amount of folate received from food intake or what is usually taken during pregnancy) may be needed.

A randomized controlled trial was conducted in 70 obstetrical centres in 5 countries (Argentina, Australia, Canada, Jamaica, and the UK) to evaluate the effect of high dose folic acid started in early pregnancy on the risk of developing preeclampsia in high-risk women. A sample size of 2464 allowed for 80% power and a 10% loss to follow-up/study withdrawal. Participants received either placebo or four 1.0 mg oral tablets of folic acid.

ELIGIBILITY:
Inclusion Criteria:

1. Capability of subject to comprehend and comply with study requirements
2. ≥ 18 years of age at time of consent
3. Subject is taking ≤1.1 mg of folic acid daily at the time of randomization
4. Live fetus (documented positive fetal heart prior to randomization)
5. Gestational age between 8+0 and 16+6 weeks of pregnancy (Gestational age (GA) of subjects will be calculated based on the first day of the last menstrual period (LMP) or ultrasound performed before 12+6. If early ultrasound and LMP dates differ by ≤ 7 days, base GA estimate on LMP date; if > 7 days, use early < 12+6 ultrasound)
6. Subject plans to give birth in a participating hospital site
7. Pregnant subjects must fulfill at least one of the following identified risk factors for pre-eclampsia (PE):

   * Pre-existing hypertension (documented evidence of diastolic blood pressure ≥ 90 mmHg on two separate occasions or at least 4 hours apart prior to randomization, or use of antihypertensive medication during this pregnancy specifically for the treatment of hypertension prior to randomization)
   * Pre-pregnancy diabetes (documented evidence of Type I or type II DM)
   * Twin pregnancy
   * Documented evidence of history of PE in a previous pregnancy
   * BMI > 35 kg/m2 within 3 months prior to this pregnancy and up to randomization of this pregnancy (documented evidence of height and weight to calculate BMI is required)

Exclusion Criteria:

1. Known history or presence of any clinically significant disease or condition which would be a contraindication to folic acid supplementation of up to 5 mg daily for the duration of pregnancy
2. Known major fetal anomaly or fetal demise
3. History of medical complications, including:

   * renal disease with altered renal function,
   * epilepsy,
   * cancer, or
   * use of folic acid antagonists such as valproic acid
4. Individual who is currently enrolled or has participated in another clinical trial or who received an investigational drug within 3 months of the date of randomization (unless approved by the Trial Coordinating Centre)
5. Known presence of:

   * Alcohol abuse (≥ 2 drinks per day) or alcohol dependence
   * Illicit drug/substance use and/or dependence
6. Known hypersensitivity to folic acid
7. Multiple Pregnancy (triplets or more)
8. Participation in this study in a previous pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2464 (Actual)
Dates: Start 2011-04; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shi Wu Wen, PhD, Principal Investigator — Ottawa Hospital Research Institute; Mark C Walker, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (72):
- Argentina (8):
  - Hospital Escuela Eva Perón, Rosario, Santa Fe Province
  - Hospital Provincial, Rosario, Santa Fe Province
  - Hospital Roque Saenz Penia, Rosario, Santa Fe Province
  - Maternidad Martin, Rosario, Santa Fe Province
  - Sanatorio de la Mujer, Rosario, Santa Fe Province
  - Cemic, Buenos Aires
  - Hospital Cullen, Santa Fe
  - Hosptial Iturraspe, Santa Fe
- Australia (6):
  - Nepean, Penrith, New South Wales
  - Townsville, Douglas, Queensland
  - Ipswich, Ipswich, Queensland
  - Adelaide, North Adelaide, South Australia
  - Royal Women's Hospital, Parkville, Victoria
  - Sunshine, St Albans, Victoria
- Canada (23):
  - Calgary Foothills Medical Center, Calgary, Alberta
  - Edmonton Lois Hole Hospital for Women, Edmonton, Alberta
  - Vancouver BC Women's Hospital and Health Center, Vancouver, British Columbia
  - St-Paul's Hospital, Vancouver, British Columbia
  - Fredericton Dr. Everett Chalmers Regional Hospital, Fredericton, New Brunswick
  - Moncton Hospital, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Winnipeg St. Boniface General Hospital, Winnipeg, New Brunswick
  - Winnipeg University of Manitoba, Winnipeg, New Brunswick
  - St-John's Women's Health Centre, St. John's, Newfoundland and Labrador
  - Hamilton McMaster University, Hamilton, Ontario
  - Kingston, Kingston, Ontario
  - London, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Civic Hospital, Ottawa, Ontario
  - Sault Ste- Marie Sault Area Hospital, Sault Ste. Marie, Ontario
  - Sunnybrook Health Sciences, Toronto, Ontario
  - Quebec City (CHUL) Centre Hospitalier Universitaire, Montreal, Quebec
  - Saint-Luc CHUM - Montreal, Montreal, Quebec
  - McGill University Royal Victoria Hospital, Montreal, Quebec
  - Sainte-Justine, Montreal, Quebec
  - St-Mary's Hospital, Montreal, Quebec
  - Regina Qu'Appelle Health Region, Regina, Saskatchewan
- Jamaica (3):
  - Jubilee, Kingston
  - Spanishtown, Kingston
  - University of West Indies, Kingston
- United Kingdom (32):
  - Hinchingbrooke, Huntingdon, Cambridgeshire
  - Warrington and Halton Hospitals NHS Foundation Trust, Warrington, Cheshire
  - Darlington Memorial Hospital, Darlington, County Durham
  - University Hospital of North Durham, Durham, County Durham
  - Cumberland Infirmary, Carlisle, Cumbria
  - West Cumberland Hospital, Whitehaven, Cumbria
  - Fairfield, Bury, Lancashire
  - Rochdale, Rochdale, Lancashire
  - Lincolnshire, Lincoln, Lincolnshire
  - Ormskirk, Southport, Merseyside
  - Northwick Park Hospital, Harrow, Middlesex
  - West Middlesex University Hospital, Isleworth, Middlesex
  - 49 Marine Avenue & CCGs, Whitley Bay, Newcastle Upon Tyne
  - Wansbeck General Hospital, Ashington, Northumberland
  - St George's Hospital, London, Tooting
  - Gateshead Queen Elizabeth Hospital, Gateshead, Tyne and Wear
  - South Tyneside District Hospital, South Shields, Tyne and Wear
  - The Royal Wolverhampton NHS Trust, New Cross Hospital, Wolverhampton, West Midlands
  - Blackburn, Blackburn
  - Burnley, Burnley
  - North Manchester, Crumpsall
  - Guy's & St Thomas' Hospital, London
  - South Tees Hospital, Middlesbrough
  - Newcastle upon Tyne Hospitals, Newcastle upon Tyne
  - North Tyneside General Hospital, North Shields
  - Norfolk & Norwich, Norwich
  - Nottingham City Hospital, Nottingham
  - Nottingham Queens Medical Centre, Nottingham
  - Oldham, Oldham
  - North Tees Hospital, Stockton
  - Sunderland Royal Hospital, Sunderland
  - Hillingdon Hospital, Uxbridge

REFERENCES:
- [Derived] Muldoon KA, McLean C, El-Chaar D, Corsi DJ, Rybak N, Dagvadorj A, Guo Y, Rennicks White R, Dingwall-Harvey ALJ, Gaudet LM, Walker MC, Wen SW; FACT Collaborating Group. Persisting risk factors for preeclampsia among high-risk pregnancies already using prophylactic aspirin: a multi-country retrospective investigation. J Matern Fetal Neonatal Med. 2023 Dec;36(1):2200879. doi: 10.1080/14767058.2023.2200879. PMID 37073421
- [Derived] Rose EG, Murphy MSQ, Erwin E, Muldoon KA, Harvey ALJ, Rennicks White R, MacFarlane AJ, Wen SW, Walker MC. Gestational Folate and Folic Acid Intake among Women in Canada at Higher Risk of Pre-Eclampsia. J Nutr. 2021 Jul 1;151(7):1976-1982. doi: 10.1093/jn/nxab063. PMID 33851221
- [Derived] Corsi DJ, Gaudet LM, El-Chaar D, White RR, Rybak N, Harvey A, Muldoon K, Wen SW, Walker M. Effect of high-dose folic acid supplementation on the prevention of preeclampsia in twin pregnancy. J Matern Fetal Neonatal Med. 2022 Feb;35(3):503-508. doi: 10.1080/14767058.2020.1725882. Epub 2020 Feb 18. PMID 32067533
- [Derived] Wen SW, White RR, Rybak N, Gaudet LM, Robson S, Hague W, Simms-Stewart D, Carroli G, Smith G, Fraser WD, Wells G, Davidge ST, Kingdom J, Coyle D, Fergusson D, Corsi DJ, Champagne J, Sabri E, Ramsay T, Mol BWJ, Oudijk MA, Walker MC; FACT Collaborating Group. Effect of high dose folic acid supplementation in pregnancy on pre-eclampsia (FACT): double blind, phase III, randomised controlled, international, multicentre trial. BMJ. 2018 Sep 12;362:k3478. doi: 10.1136/bmj.k3478. PMID 30209050
- [Derived] Wen SW, Champagne J, Rennicks White R, Coyle D, Fraser W, Smith G, Fergusson D, Walker MC. Effect of folic acid supplementation in pregnancy on preeclampsia: the folic acid clinical trial study. J Pregnancy. 2013;2013:294312. doi: 10.1155/2013/294312. Epub 2013 Nov 18. PMID 24349782

RESULTS

PARTICIPANT FLOW:
Recruitment Details: High risk pregnant women were recruited in Canada and internationally.
Period: Overall Study
Arm/Group | Folic Acid 4 mg | Placebo
Started | 1228 | 1236
Completed | 1144 | 1157
Not Completed | 84 | 79
Not completed — Withdrew consent | 39 | 47
Not completed — No primary outcome data | 17 | 11
Not completed — Spontaneous abortion (<20 weeks) | 22 | 15
Not completed — Early intrauterine fetal death | 6 | 6

BASELINE CHARACTERISTICS:
Population: One participant (in the Folic Acid group) withdrew consent on the same day of randomization and was excluded completely from the baseline and outcome analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Folic Acid 4 mg | Placebo | Total
Number analyzed (Participants) | 1227 | 1236 | 2463
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (5.4) | 31 (5.4) | 31 (5.4)
Age, Customized [Count of Participants; unit: Participants]
  Maternal age (years): <20 | 10 | 10 | 20
  Maternal age (years): 20-29 | 439 | 447 | 886
  Maternal age (years): 30-34 | 411 | 441 | 852
  Maternal age (years): >=35 | 367 | 338 | 705
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1227 | 1236 | 2463
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Maternal Background: Native/Aboriginal | 35 | 24 | 59
  Maternal Background: Caucasian | 970 | 987 | 1957
  Maternal Background: Black | 93 | 107 | 200
  Maternal Background: Asian | 45 | 50 | 95
  Maternal Background: Latino/Hispanic | 31 | 22 | 53
  Maternal Background: Indian/South Asian | 45 | 36 | 81
  Maternal Background: Declined to answer | 8 | 10 | 18
Region of Enrollment [Number; unit: participants]
  Canada | 600 | 607 | 1207
  Argentina | 157 | 153 | 310
  United Kingdom | 61 | 61 | 122
  Australia | 29 | 32 | 61
  Jamaica | 380 | 383 | 763
Parity [Count of Participants; unit: Participants]
  0 | 413 | 420 | 833
  1 | 498 | 499 | 997
  >=2 | 316 | 317 | 633
Pre-pregnancy BMI (kg/m2) [Count of Participants; unit: Participants]
  <18.5 | 15 | 11 | 26
  18.5 to <25 | 230 | 225 | 455
  25 to <30 | 211 | 199 | 410
  30 to <35 | 164 | 146 | 310
  >=35 | 607 | 655 | 1262
Education level [Count of Participants; unit: Participants] — 3 participants were missing education (1 in the intervention arm and 2 in the placebo arm). Therefore, only 1226 participants in the intervention arm and 1234 participants in the placebo arm had data for this baseline measure.
  Participants
    High school and below | 353 | 348 | 701
    College/University not complete | 198 | 197 | 395
    College/University completed | 675 | 689 | 1364
Gestational age (weeks) at recruitment [Count of Participants; unit: Participants]
  8-12 | 386 | 433 | 819
  13-16 | 841 | 803 | 1644
Smoking during pregnancy [Count of Participants; unit: Participants]
  Yes | 98 | 95 | 193
  No | 1046 | 1035 | 2081
  Quit during pregnancy | 83 | 106 | 189
Alcohol during pregnancy [Count of Participants; unit: Participants]
  Yes | 23 | 27 | 50
  No | 977 | 955 | 1932
  Quit during pregnancy | 227 | 254 | 481
Supplementation of FA at randomisation (yes) [Count of Participants; unit: Participants] | 989 | 1016 | 2005
Supplementation of high dose FA at randomisation (yes) [Count of Participants; unit: Participants] | 346 | 335 | 681
Aspirin supplementation at randomisation [Count of Participants; unit: Participants] | 358 | 340 | 698
Calcium supplementation at randomisation [Count of Participants; unit: Participants] | 97 | 109 | 206
Dietary Folate (µg) (Mean, SD) [Mean (Standard Deviation); unit: µg] — Dietary folate was measured at both Visit 1 and Visit 2 in the study to capture folate intake from food throughout pregnancy. Population: Remaining participants did not return study treatment and so the mean could not be calculated.
  µg
    VIsit 1 (8-16 completed weeks' gestation): number analyzed (Participants) | 1215 | 1225 | 2440
    VIsit 1 (8-16 completed weeks' gestation) | 494 (209) | 504 (222) | 499 (216)
    Visit 2 (24-26 weeks' completed gestation): number analyzed (Participants) | 1008 | 1023 | 2031
    Visit 2 (24-26 weeks' completed gestation) | 494 (209) | 500 (213) | 497 (211)
Visit 2 Compliance [Count of Participants; unit: Participants] — Participants completed the Food Frequency Questionnaire at Visit 2 to capture dietary folate during mid-pregnancy. Population: Calculated on returned study treatment (n=1941). Remaining participants did not return any study treatment and compliance could not be calculated (n=522).
  Participants
    number analyzed (Participants) | 964 | 977 | 1941
    ≤50% | 108 | 106 | 214
    50-75% | 140 | 122 | 262
    ≥75% | 716 | 749 | 1465
History of Pre-eclampsia [Count of Participants; unit: Participants] | 308 | 303 | 611
Chronic Hypertension [Count of Participants; unit: Participants] | 203 | 241 | 444
Type 1 Diabetes [Count of Participants; unit: Participants] | 84 | 72 | 156
Type 2 Diabetes [Count of Participants; unit: Participants] | 98 | 84 | 182
Twin Pregnancy [Count of Participants; unit: Participants] | 233 | 229 | 462
Body mass index >=35 [Count of Participants; unit: Participants] | 606 | 656 | 1262
Prepregnancy Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 34 (8.6) | 34 (13) | 34 (11)
Gestational age at recruitment [Mean (Standard Deviation); unit: weeks] | 14 (1.9) | 14 (1.9) | 14 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Preeclampsia
Description: PE is defined as diastolic blood pressure ≥90 mmHg on two occasions ≥4 hours apart and proteinuria developed in women greater than 20+0 weeks of gestation. Proteinuria is defined as: urinary protein ≥300mg in 24 hour urine collection OR in the absence of 24 hour collection, ≥2+ dipstick proteinuria, OR random protein-creatinine ratio ≥30mg protein/mmol.
  OR HELLP (Haemolysis, Elevated, Liver Enzymes, Low Platelets) syndrome defined as: Haemolysis (characteristic peripheral blood smear), Serum LDH ≥ 600U/L, Serum AST ≥ 70U/L, and Platelet count <100 x109/L
  OR Superimposed pre-eclampsia, defined as history of pre-existing hypertension (diagnosed pre-pregnancy or before 20+0 weeks' gestation) with new proteinuria.
Time Frame: Participants will be followed from 20+0 weeks of gestational age until 42 days postpartum (after delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1144 | 1157
Participants | 169 | 156
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.37, Chi-squared; Risk Ratio (RR) = 1.10, 95% CI 2-sided [0.90 to 1.34]

2. Secondary Outcome: Maternal Death
Description: According to the World Health Organization, "A maternal death is defined as the death of a woman while pregnant or within 42 days of termination of pregnancy, irrespective of the duration and site of the pregnancy, from any cause related to or aggravated by the pregnancy or its management but not from accidental or incidental causes.
Time Frame: Time Frame: Participants will be followed from 20+0 weeks of gestation until 42 days postpartum (after delivery)
Population: Participants who completed study and were analyzed for primary outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1144 | 1157
Participants | 0 | 0

3. Secondary Outcome: Spontaneous Abortion
Description: Spontaneous abortion or miscarriage defined as death of a fetus <500g or <20 weeks of gestation
Time Frame: Participants will be followed from randomization until 20+0 weeks of gestation
Population: Not all participants had secondary outcome data. Numbers above reflect those that had information available for this secondary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1172 | 1180
Participants | 27 | 21
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.37, Chi-squared; Risk Ratio (RR) = 1.29, 95% CI 2-sided [0.74 to 2.28]

4. Secondary Outcome: Placenta Abruption
Description: Placental abruption (abruptio placentae) is the premature detachment of a normally positioned placenta from the wall of the uterus.
Time Frame: Participants will be followed from 20+0 weeks of gestation until delivery
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1169 | 1179
Participants | 12 | 19
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.21, Chi-squared; Risk Ratio (RR) = 0.64, 95% CI 2-sided [0.31 to 1.31]

5. Secondary Outcome: Premature Rupture of Membranes
Description: Rupture of the membranes (rupture of the amniotic sac) before the onset of labor.
Time Frame: Participants will be followed from randomization (8-16 weeks' completed gestation) until the onset of labor
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1169 | 1180
Participants | 215 | 224
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.71, Chi-squared; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.82 to 1.15]

6. Secondary Outcome: Preterm Birth
Description: Birth that occur earlier than 37+0 weeks of gestational age.
Time Frame: Participants will be followed from 20+0 weeks to 36+6 weeks of gestation
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1150 | 1164
Participants | 297 | 304
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.87, Chi-squared; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.86 to 1.13]

7. Secondary Outcome: HELLP (Hemolysis, Elevated Liver Enzyme Levels & Low Platelet Count)
Description: Haemolysis (characteristic peripheral blood smear), Serum LDH >=600U/L, Serum AST >=70U/L, Platelet count <100 x109/L
Time Frame: Participants will be followed from 20+0 weeks of gestation until delivery
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1144 | 1156
Participants | 6 | 5
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.75, Chi-squared; Risk Ratio (RR) = 1.21, 95% CI 2-sided [0.37 to 3.96]

8. Secondary Outcome: Severe Preeclampsia
Description: Severe PE: Defined as PE with convulsion or HELLP or delivery <34 weeks.
Time Frame: Participants will be followed from 20+0 weeks of gestation until delivery.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1144 | 1156
Participants | 24 | 16
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.19, Chi-squared; Risk Ratio (RR) = 1.52, 95% CI 2-sided [0.81 to 2.84]

9. Secondary Outcome: Antenatal Inpatient Length of Stay
Description: Length of inpatient stay before admission for delivery in days
Time Frame: Participants will be followed from date of randomization (8-16 weeks' completed gestation) until admission for delivery
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 221 | 232
days | 5.6 (7.7) | 5.2 (6.2)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.61, t-test, 2 sided; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-0.96 to 1.63], Standard Deviation 7.0

10. Secondary Outcome: Stillbirth
Description: Fetal death defined as death of fetus of at least 500 grams birth weight or, if birth weight is unavailable, a gestational age of at least 20+0 weeks of gestation.
Time Frame: Participants will be followed from 20+0 weeks of gestation up to delivery.
Population: A total of 2738 infants were born to women recruited into the trial (1364 in folic acid group and 1374 in placebo group). This is an infant outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1364 | 1374
Participants | 15 | 26
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.14, Chi-squared; Risk Ratio (RR) = 0.60, 95% CI 2-sided [0.30 to 1.19]

11. Secondary Outcome: Intrauterine Growth Restriction (<3rd Percentile)
Description: Intrauterine growth restriction is defined as a birth weight less than the 3rd percentile of the population, adjusted for sex and gestational age, based on the current population-based Canadian reference standard.
Time Frame: Participants will be followed from 20+0 weeks of gestation until delivery
Population: A total of 2738 infants were born to women recruited into the trial (1364 in folic acid group and 1374 in placebo group). This is an infant outcome. Some participants had missing data for this outcome and therefore were excluded from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1347 | 1348
Participants | 20 | 25
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.37, Chi-squared; Risk Ratio (RR) = 0.76, 95% CI 2-sided [0.41 to 1.39]

12. Secondary Outcome: Intrauterine Growth Restriction (<10th Percentile)
Description: Intrauterine growth restriction is defined as a birth weight less than the 10th percentile of the population, adjusted for sex and gestational age, based on the current population-based Canadian reference standard.
Time Frame: Participants will be followed from 20+0 weeks of gestation until delivery
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1347 | 1348
Participants | 151 | 144
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.82, Chi-squared; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.81 to 1.30]

13. Secondary Outcome: Neonatal Death
Description: Neonatal death defined as death of a baby that occurred during first 28 days of life.
Time Frame: Participants will be followed from birth until 28 days of life
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1343 | 1347
Participants | 8 | 11
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.79, Chi-squared; Risk Ratio (RR) = 0.87, 95% CI 2-sided [0.31 to 2.44]

14. Secondary Outcome: Perinatal Mortality
Description: The perinatal mortality is defined as the number of deaths (fetal deaths and neonatal deaths) of babies ≥ 500 grams birth weight or, if birth weight is unavailable, a gestational age ≥ 20+0 weeks, up to 28 completed days after birth.
Time Frame: Participants will be followed from 20+0 weeks of gestation until 28 days of life.
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1364 | 1374
Participants | 23 | 37
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.07, Chi-squared; Risk Ratio (RR) = 0.63, 95% CI 2-sided [0.37 to 1.05]

15. Secondary Outcome: Retinopathy of Prematurity
Description: Retinopathy of prematurity a retinopathy typically occurring in premature infants treated with high concentrations of oxygen, characterized by vascular dilatation, proliferation, tortuosity, edema, retinal detachment, and fibrous tissue behind the lens confirmed by retinal examination according to an International Committee for the Classification of Retinopathy of Prematurity.
Time Frame: Infants born to the participant will be followed for the duration of hospital stay, or up to 6 weeks
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1342 | 1347
Participants | 21 | 13
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.65, Chi-squared; Risk Ratio (RR) = 1.20, 95% CI 2-sided [0.54 to 2.66]

16. Secondary Outcome: Early Onset Sepsis
Description: Within first 48hr of life, confirmed by positive blood or cerebrospinal fluid cultures
Time Frame: Infants born to the participants will be followed first 48 hours of life.
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1342 | 1347
Participants | 3 | 9
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.10, Chi-squared; Risk Ratio (RR) = 0.34, 95% CI 2-sided [0.09 to 1.23]

17. Secondary Outcome: Necrotising Enterocolitis
Description: Necrotizing enterocolitis (NEC) according to modified Bell's criteria stage 2 or higher (grossly bloody stool, plus absent bowel sounds with or without abdominal tenderness and radiographic findings such as intestinal dilation, ileus, pneumatosis intestinalis), excluding isolated spontaneous intestinal perforations.
Time Frame: Infants borm to the participants will be followed for the duration of hospital stay, or up to 6 weeks.
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1343 | 1347
Participants | 8 | 3
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.33, Chi-squared; Risk Ratio (RR) = 2.04, 95% CI 2-sided [0.49 to 8.57]

18. Secondary Outcome: Intraventricular Hemorrhage (IVH)
Description: * IVH Grade 1(Blood in germinal matrix)
  * IVH Grade 2 (Blood in germinal matrix and extending into the ventricles)
  * IVH Grade 3 (Ventricular enlargement)
  * IVH Grade 4 (Intraparenchymal lesion)
Time Frame: Time Frame: Infants born to the participants will be followed for the duration of hospital stay, or up to 6 weeks
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1343 | 1347
Participants | 18 | 19
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.94, Chi-squared; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.47 to 2.00]

19. Secondary Outcome: Ventilation
Description: Ventilatory support after initial resuscitation, with/without intubation.
Time Frame: Infants born to the participants will be followed for the duration of hospital stay, or up to 6 weeks.
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1346 | 1348
Participants | 49 | 30
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.06, Chi-squared; Risk Ratio (RR) = 1.61, 95% CI 2-sided [0.97 to 2.66]

20. Secondary Outcome: Need for Oxygen at 28 Days
Time Frame: Infants to the participants will be followed for 28 days after birth.
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1220 | 1227
Participants | 9 | 3
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.21, Chi-squared; Risk Ratio (RR) = 2.37, 95% CI 2-sided [0.61 to 9.14]

21. Secondary Outcome: Composite Severe Adverse Fetal/Neonatal Outcome
Description: Composite outcome included any of retinopathy of prematurity, periventricular leukomacia, early onset sepsis, necrotizing enterocolitis, intraventricular haemorrhage, ventilation. Need for O2at 28 days, NICU admission
Time Frame: Outcomes included in the composite outcome were measured for each of their respective time frames, up to 6-weeks after birth
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1349 | 1348
Participants | 63 | 51
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.38, Chi-squared; Risk Ratio (RR) = 1.20, 95% CI 2-sided [0.80 to 1.80]

22. Secondary Outcome: Length of Stay in 'High Level' Neonatal Care Unit
Time Frame: Infants to the participants will be followed for the duration of hospital stay, or up to 6 weeks.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 299 | 263
days | 16 (27) | 17 (23)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 046, t-test, 2 sided; Mean Difference (Net) = -1.60, 95% CI 2-sided [-5.84 to 2.64]

23. Secondary Outcome: Neonatal Death
Description: Neonatal death defined as death of the infant occurred before 28 days of life
Time Frame: Infants to the participants will be followed for 28 days after birth.
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1343 | 1347
Participants | 151 | 144
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.79, Chi-squared; Risk Ratio (RR) = 0.87, 95% CI 2-sided [0.31 to 2.44]

24. Secondary Outcome: Periventricular Leukomalacia
Description: One of the two outcomes used to measure neonatal morbidity.
Time Frame: Infants to the participants were followed for 28 days after birth.
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1343 | 1347
Participants | 4 | 2
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.42, Chi-squared; Risk Ratio (RR) = 2.00, 95% CI 2-sided [0.37 to 10.92]

25. Secondary Outcome: Neonatal Intensive Care Unit (NICU) Admission
Description: This outcome measured whether or not the infant was admitted into the NICU.
Time Frame: Infants to the participants will be followed for the duration of hospital stay, or up to 6 weeks.
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid 4 mg | Placebo
Number analyzed (Participants) | 1346 | 1348
Participants | 299 | 267

ADVERSE EVENTS:
Description: One participant (in the Folic Acid group) withdrew consent on the same day of randomization; participants is excluded from being considered "at risk" for AE/SAEs.
Arm/Group | Folic Acid 4 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 227/1227 | 195/1236
Other Adverse Events (participants affected / at risk) | 961/1227 | 968/1236
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Folic Acid 4 mg (N=1227) | Placebo (N=1236)
Prematurity (Pregnancy, puerperium and perinatal conditions) | 29 | 20
Hypertension (Pregnancy, puerperium and perinatal conditions) | 31 | 25
Other SAE (Pregnancy, puerperium and perinatal conditions) | 167 | 150
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Folic Acid 4 mg (N=1227) | Placebo (N=1236)
Other AE (Pregnancy, puerperium and perinatal conditions) | 961 | 968

LIMITATIONS AND CAVEATS:
The diagnosis of PE is complex due to its heterogenous aetiology. The criteria for PE have remained consistent with NICE guidelines, but there have been revisions in other settings. Therefore additional women in the study might have had PE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes